CLINICAL TRIAL: NCT07257094
Title: French Validation of the Nasal Reconstruction FACE-Q Questionnaire for Reconstruction/Rehabilitation Following Nasal Skin Cancer
Brief Title: Nasal Reconstruction FACE-Q : French Validation of the Nasal Reconstruction FACE-Q Questionnaire for Reconstruction/Rehabilitation Following Nasal Skin Cancer
Status: Recruiting | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-A02195-44; CHRD 1424 (Other: HOPITAL NOVO)
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma
Keywords: Basal Cell carcinoma; Squamous Cell carcinoma; Rhinectomy; Reconstructive Surgical Procedures; Prosthesis Implantation; FACE-Q; Quality of Life
MeSH Terms: conditions — Carcinoma; Carcinoma, Basal Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Operated patients: Patients with skin cancer in the nasal region who have undergone surgical reconstruction using a flap or rehabilitation using a prosthesis.
  Interventions: Other: operated patients
- Control: Patients with no history of surgery or facial trauma
  Interventions: Other: Control

INTERVENTIONS:
Other: operated patients — Response to the Nasal Reconstruction FACE-Q questionnaire, which includes the following scales :
  * Appearence : Face overall, nose, nostrils, skin
  * Health related quality of life (HRQOL) : Early life impact, psychological, social, outcome
  * Adverse effects : on the nose, on the forehead, eyebrows and scalp
  * Nasal Obstruction Symptom Evaluation (NOSE)
  * Short-Form-36 (SF 36)
  Groups: Operated patients
Other: Control — Response to the Nasal Reconstruction FACE-Q questionnaire, which includes the following scales :
  * Appearence : Face overall, nose, nostrils, skin impact psychological, impact social,
  * SF36
  Groups: Control

SUMMARY:
This study aims to validate a French version of the Nasal Reconstruction FACE-Q questionnaire for patients who have undergone nasal reconstruction or prosthetic rehabilitation after surgery for nasal skin cancer. The questionnaire evaluates appearance, quality of life, and possible side effects related to the reconstruction.

The investigators hypothesize that the validated French version will provide a reliable and standardized tool to assess patient satisfaction and health-related quality of life in this context.

DETAILED DESCRIPTION:
Nasal skin cancers often require surgical excision that can result in significant tissue loss. Treatment may involve complex surgical reconstruction or, in some cases, prosthetic rehabilitation. These procedures may have major aesthetic, functional, and psychological consequences.

FACE-Q is an internationally recognized, patient-reported outcome instrument designed to assess satisfaction with appearance, health-related quality of life, and treatment-related adverse effects. However, FACE-Q was developed and validated in English and requires cultural and linguistic adaptation for reliable use in French-speaking populations.

This non-interventional, multicenter study aims to translate and validate the relevant FACE-Q Aesthetics scales in French for patients who have undergone nasal reconstruction or prosthetic rehabilitation after skin cancer. The selected domains address facial and nasal appearance, psychosocial well-being, social function, satisfaction with outcomes, and procedure-related adverse effects.

The expected outcome is to provide a standardized and validated French-language tool that reliably evaluates these patients' satisfaction and quality of life. Such a tool may be applied in clinical practice and future comparative research to improve patient care.

ELIGIBILITY:
PATIENTS

Inclusion Criteria

* Age ≥ 18 years
* Patient who has undergone excision of a cutaneous, mucocutaneous, or vestibular nasal cancer with surgical reconstruction using a flap or prosthetic rehabilitation, performed more than 4 months ago, with stable results, and less than 3 years ago
* Patient informed of the study and not opposed to participation

Exclusion Criteria

* Patient under anticoagulant or antiplatelet therapy Non-French-speaking patient
* Patient under legal protection (e.g., guardianship, legal safeguard) or with limited legal capacity
* Patient unlikely to cooperate with the study and/or poor anticipated compliance as judged by the investigator (including psychiatric disorders other than depressive disorder or cognitive impairment)
* Pregnant or breastfeeding woman

CONTROL

Inclusion Criteria

* Age ≥ 65 years
* Subject informed and not opposed to participating in the study
* Subject who has never undergone facial trauma or surgery, and without major comorbidity, defined as follows:
* No heart failure (moderate or severe heart failure, history of heart attack within the last 6 months);
* No severe chronic respiratory disease (no stage III-IV COPD, no prolonged oxygen therapy);
* No uncontrolled diabetes or associated severe complications;
* No active immunosuppressive diseases or high-dose immunosuppressive treatment;
* No unstable or severe facial dermatological conditions;
* No comorbidities seriously affecting quality of life or respiratory function (at the investigator's discretion).

Exclusion Criteria

* Non-English speaking subject
* Subject under guardianship or legal protection, legally incompetent or with limited legal capacity
* Subject unlikely to cooperate in the study and/or anticipated low cooperation by the investigator (particularly those with psychiatric disorders other than depression or cognitive disorders)
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients / Controls
Sampling Method: Non-Probability Sample
Enrollment: 346 (Estimated)
Dates: Start 2026-01-10 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Psychometric validation of the French version of Nasal Reconstruction FACE-Q | 7 days
  Test the acceptability, reliability, construct validity, and sensitivity to change of the questionnaire.

SECONDARY OUTCOMES:
Assessment of the post operative functional satisfaction | 7 days
  Evaluation of postoperative functional satisfaction using the Nasal Obstruction Symptom Evaluation (NOSE) questionnaire, which measures the severity of nasal breathing obstruction. Correlations will then be calculated between the NOSE score and each of the FACE-Q scales.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled AL TABAA, Doctor, Study Director — Hôpital NOVO
Locations (9):
- France (9):
  - CHU Caen, Caen
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Hôpital Lariboisière (AP-HP), Paris
  - Hôpital Bichat (APHP), Paris
  - Hopital Novo, Pontoise
  - HNIA Toulon, Toulon
  - CHU Toulouse, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No